CLINICAL TRIAL: NCT01969656
Title: A Phase 1B, Double-Blind, Placebo-Controlled, Calcitriol Active-Controlled, Daily-Dose, Escalating-Dose, Safety and Tolerance Study of 2MD Soft Gel Capsules in Normal Healthy Postmenopausal Women
Brief Title: Safety Study of an Oral Vitamin D Analog in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deltanoid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2MD-3H-1B/C
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Postmenopausal Osteoporosis, Multiple Sites
Keywords: vitamin D analog
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Calcitriol

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Calcitriol (Active Comparator)
  Interventions: Drug: Calcitriol
- 50 ng 2MD (Experimental)
  Interventions: Drug: 2MD
- 110 ng 2MD (Experimental)
  Interventions: Drug: 2MD
- 170 ng 2MD (Experimental)
  Interventions: Drug: 2MD
- 220 ng 2MD (Experimental)
  Interventions: Drug: 2MD
- 440 ng 2MD (Experimental)
  Interventions: Drug: 2MD

INTERVENTIONS:
Drug: 2MD
  Arms: 110 ng 2MD; 170 ng 2MD; 220 ng 2MD; 440 ng 2MD; 50 ng 2MD
Drug: Calcitriol
  Arms: Calcitriol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Determine the safety of 2MD, a vitamin D analog, when administered orally once daily for 28 days in healthy normal postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy postmenopausal women, ≥ 60 but ≤ 80 years of age, or between 45 and 60 years of age who have been amenorrheic for at least 2 years plus have a serum FSH level of > 30 IU/L, or women with a documented bilateral oophorectomy at least 2 years prior to study start.
2. Within ±30% of their ideal body weight for height and body frame.
3. Demonstrated ability to understand and willingness to sign an Informed Consent Form.
4. 24-hour urinary Ca ≤250 mg/day and a urinary Ca:Cr ≤0.35.
5. Negative urine test for selected drugs of abuse.
6. Willing to maintain a total calcium intake between 700 and 1000 mg/day.

Exclusion Criteria:

1. Any acute or chronic condition that would limit the subject's ability to complete the study.
2. Active clinical manifestations of significant metabolic, hematological, pulmonary, hepatic, cardiovascular, gastrointestinal (including malabsorption), neurological, renal, urological or psychiatric disorders.
3. History or presence of any diseases known or believed to influence calcium absorption or metabolism.
4. History of renal calculi.
5. History of an eating disorder.
6. History of stomach or intestinal surgery.
7. History of hypersensitivity or allergies to any vitamin D derivative.
8. History or presence of an abnormal ECG.
9. Use of any medications or products affecting vitamin D metabolism within 6 months prior to study entry.
10. Use of any medications or products affecting calcium balance or bone turnover within 6 months prior to study entry.
11. Participation in any other investigational study drug trial in which receipt of investigational study drug occurred within 60 days prior to study entry.
12. Use of vitamin and/or mineral supplements >1X RDI within 4 weeks prior to study entry, unless deemed acceptable by Investigator.
13. Poor peripheral venous access.
14. Receipt of blood products within 2 months prior to study entry.

    -

Ages: 45 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total serum calcium | Days 0 (pre-dose), 1, 2, 3, 7, 14, 21, 27, 28 and 2 weeks after last dose
Change from baseline in levels of 2MD in the blood | 1, 2, 3, 12, 18 and 24 h after the initial dose on Day 0 and after the final dose on Day 27